CLINICAL TRIAL: NCT05343416
Title: NaROA STUDY: OBSERVATIONAL, PROSPECTIVE, MULTICENTRIC, NATIONAL OPEN ABDOMEN REGISTRY FOR THE ANALYSIS OF INDICATIONS AND PRONOTIC FACTORS OF MORBI-MORTALITY IN PATIENTS UNDERGOING EMERGENCY SURGERY BY GENERAL SURGERY.
Brief Title: NaROA STUDY: National Register of Open Abdomen
Acronym: NaROA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Amalia Pelegrina, Principal Investigator, Hospital del Mar
Other Study IDs: Register of Open Abdom
Record Dates: First submitted 2021-02-23; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-01

CONDITIONS: Open Abdomen Technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open abdomen procedure: All patients underwent to open abdomen procedure
  Interventions: Procedure: Open abdomen procedure

INTERVENTIONS:
Procedure: Open abdomen procedure — All patients underwent to open abdomen procedure

SUMMARY:
National Register of Open Abdomen Open Abdomen Procedure (Observational and Prospective Study)

DETAILED DESCRIPTION:
The open abdomen technique has widely been proven useful in the treatment of traumatic patients, but its indication in non-traumatic patients with catastrophic abdomen (peritonitis, ischaemia, pancreatitis) generates controversy. Its heterogeneous implementation is based on insufficient evidence and originated in health systems very different from ours. Its low prevalence imposes the need for a multicentre study.

AIMS : Establish a national, prospective, multi-centre national registry of non traumatic patients with open abdominal indication whether or not they undergo damage control surgery and open abdomen for:

1. Describe in real time the indications, surgical technique, materials, time, risk factors, definitive closure, reinterventions and complications according to the Clavien-Dindo classification and mortality.
2. Compare the results of the application or non-application of the open abdomen in non-traumatic patients between the different participating centers.
3. Set the limits of the open abdomen in non-traumatic patients indication.

ELIGIBILITY:
Inclusion Criteria:

* Indication to Open Abdomen in non-trauma patients
* Informed consent

Exclusion Criteria:

* Open Abdomen in trauma patients
* No indication to Open Abdomen
* Informed consent refusal

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients underwent to open abdomen procedure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
OPEN ABDOMEN: NON-TRAUMATIC ABDOMINAL EMERGENCIES | two years
  The open abdomen technique has widely been proven useful in the treatment of traumatic patients, but its indication in non-traumatic patients with catastrophic abdomen (peritonitis, ischaemia, pancreatitis) generates controversy. Its heterogeneous implementation is based on insufficient evidence and originated in health systems very different from ours. Its low prevalence imposes the need for a multicentre study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari del Mar (PSMar), Barcelona, Spain